CLINICAL TRIAL: NCT04528927
Title: Evaluation of the Efficacy and Safety of Treatments for Patients Hospitalized for COVID-19 Infection Without Signs of Acute Respiratory Failure, in Tunisia Multicentric Randomized Comparative Study
Brief Title: Evaluation of the Efficacy and Safety of Treatments for Patients Hospitalized for COVID-19 Infection Without Signs of Acute Respiratory Failure, in Tunisia
Acronym: THINC
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: - Interest in the use of HCQ is controversial.
Sponsor: Abderrahmane Mami Hospital (Other)
Collaborators: Eshmoun Clinical Research Center (Network); Datametrix (Industry)
Responsible Party: Principal Investigator, Dr Jalila Ben Khelil, Head of department, Abderrahmane Mami Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECC2020-05
Record Dates: First submitted 2020-05-06; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: COVID 19; Patients Hospitalized
MeSH Terms: conditions — COVID-19 | interventions — Azithromycin; Doxycycline; Zinc

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HCQ+Azithromycin (Experimental): * Hydroxychloroquine (HCQ): 600 mg on the 1st day as a starting dose then 200 mg * 2 / D for 9 days
  * Azithromycin: 500 mg (1st day) then 250 mg / D for 4 days
  * Usual standard treatment
  Interventions: Drug: HCQ; Drug: Azithromycin
- HCQ+Azithromycin+Zinc (Experimental): * HCQ: 600 mg on the 1st day as a starting dose then 200 mg * 2 / D for 9 days
  * Azithromycin: 500 mg (1st day) then 250 mg / D for 4 days
  * Zinc: 220 mg per day for 10 days
  * Usual standard treatment
  Interventions: Drug: HCQ; Drug: Azithromycin; Dietary Supplement: Zinc
- Azithromycin+Doxycycline (Experimental): * Azithromycin: 500 mg (1st day) then 250 mg / D for 4 days
  * Doxycycline: 200 mg per day for 10 days.
  * Usual standard treatment
  Interventions: Drug: Azithromycin; Drug: Doxycycline

INTERVENTIONS:
Drug: HCQ — 600 mg on the 1st day as a starting dose then 200 mg * 2 /D for 9 days
  Arms: HCQ+Azithromycin; HCQ+Azithromycin+Zinc
Drug: Azithromycin — 500 mg (1st day) then 250 mg / D for 4 days
Drug: Doxycycline — 200 mg per day for 10 days
  Arms: Azithromycin+Doxycycline
Dietary Supplement: Zinc — 220 mg per day for 10 days
  Arms: HCQ+Azithromycin+Zinc

SUMMARY:
Evaluation of the efficacy and safety of Treatments for Patients Hospitalized for COVID-19 Infection without signs of acute respiratory failure, in Tunisia Multicentric Randomized Comparative Study

DETAILED DESCRIPTION:
Arm 1:

* Hydroxychloroquine (HCQ): 600 mg on the 1st day as a starting dose then 200 mg * 2 /D for 9 days
* Azithromycin: 500 mg (1st day) then 250 mg / D for 4 days
* Usual standard treatment

Arm 2:

* HCQ: 600 mg on the 1st day as a starting dose then 200 mg * 2 / D for 9 days
* Azithromycin: 500 mg (1st day) then 250 mg / D for 4 days
* Zinc: 220 mg per day for 10 days
* Usual standard treatment

Arm 3:

* Azithromycin: 500 mg (1st day) then 250 mg / D for 4 days
* Doxycycline: 200 mg per day for 10 days.
* Usual standard treatment

ELIGIBILITY:
Inclusion Criteria:

* Confirmed patient COVID19 positive with clinical signs of acute lower respiratory infection with signs of pneumonia or bronchitis: fever and / or cough and / or difficulty breathing in the absence of acute respiratory failure (PaO2> 60 mmHg) with Plus or less :

  * Chills
  * Asthenia, fatigability
  * Headache
  * Arthromas myalgia
  * Dry throat
  * Rhinorrhea
  * An anosmia
  * chest pain
  * Diarrhea
  * Nausea and vomiting

    * Absence of rhythm disturbance (Qt interval <500ms)
    * Patients hospitalized in the medical service
    * 18 years old <Age <80 years old
    * Having given written consent for their participation in the study

Exclusion Criteria:

* Allergy to macrolides, local anesthetics such as lidocaine or amide type and betalactamines
* Take hydroxychloquine in the previous month
* Severe / severe liver failure
* Kidney failure (GFR <30 ml / min / 1.73 m2)
* Ongoing treatments with colchicine, ergot, rye, pimozide, mizolastine, simvastatin, lomitapide, alfuzosin, dapoxetine, avanafil, ivabradine, eplerenone, dronedarone, quetiapine, ticagrelor, cisapride, astemizole, terfenadine, ranolazine, domperidone.
* Complete branch block
* Hypovolemia
* Retinopathy including vitreous involvement
* Psoriasis
* Pregnant or breastfeeding woman
* hypersensitivity to chloroquine or hydroxychloroquine or to any of the other ingredients of this medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-15 (Estimated); Primary Completion 2020-07-15 (Estimated); Study Completion 2020-07-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate the rate of patients cured at the end of the study. | 2 months
  The healing criteria are defined clinically as:
  disappearance of clinical signs of acute respiratory infection absence of fever
Evaluate the rate of patients are pauci-symptomatic at the end of the study. | 2 months
  A patient will be defined as pauci-symptomatic if presence:
  * Light dry cough
  * Discomfort,
  * More or less :
    * Headache,
    * Muscle pain

SECONDARY OUTCOMES:
Evaluate the rate of patients with worsening clinical signs | 2 months
  Patients require transfer to intensive care with the appearance of:
  * Acute respiratory failure: PaO2 <60 mmHg in AA gold
  * Signs of circulatory insufficiency: mottling, tachycardia, systolic BP ≤90mmHg or having dropped by 40 mmHg compared to base BP or
  * Confusion or alteration of the state of consciousness

CONTACTS AND LOCATIONS:
Locations (1):
- Eshmoun Clinical Research Centre, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No